CLINICAL TRIAL: NCT00466986
Title: A Phase II, Non-Randomized Study of Abraxane Plus Carboplatin in Patients With Recurrent Platinum-Sensitive Ovarian or Primary Peritoneal Cancer
Brief Title: Abraxane Plus Carboplatin for Recurrent Platinum-Sensitive Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Southeastern Gynecologic Oncology (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WIRB#20051730
Record Dates: First submitted 2007-04-26; First posted 2007-04-27 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Cancer
Keywords: recurrent; ovarian; cancer; platinum sensitive
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Recurrence; Neoplasms | interventions — Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Abraxane — Carboplatin day1 every 28days. Abraxane day1,8,15 every 28days

SUMMARY:
The purpose of this study is to determine if the combination of Abraxane and Carboplatin together will improve the chances of controlling recurrent ovarian/fallopian tube/peritoneal cancer.

DETAILED DESCRIPTION:
Current best practice recommends Carboplatin combined with Taxol in the treatment of Ovarian cancer.

Taxol is paclitaxel in the solvent Cremophor-El and the solvent has been associated with significant side effects e.g. anaphylaxis and hypersensitivity. this requires the routine use of premedication with antihistamines and steroids.

Abraxane by contrast is Cremophor-El free and is protein bound. This has 2 advantages over Taxol.

1. No need for routine premedications
2. Increased drug entry into cells facilitating greater potential for anti-tumor activity.

Schedule: Carboplatin day1 every 28days. Abraxane day1,8,15 every 28days.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed recurrent epithelial ovarian or primary peritoneal carcinoma. Patient will have been staged at diagnosis according to FIGO Classification.
2. Measurable Disease by RECIST Criteria (defined by the presence of at least 1 measurable lesion (see Section 7.7.1 for definition of measurable lesions) or elevated CA-125 in the absence of measurable disease. A pre-treatment sample of CA-125 will be collected within 2 weeks before treatment is started. A pre-treatment sample of CA-125 should be at least twice the upper limit of normal.
3. Patients must have disease recurrence 6 months or more after completion of front-line platinum and paclitaxel-containing regimen. Duration of response from prior therapy and prior consolidation therapy will be documented in case report forms for descriptive analysis.
4. Patients must have received at least 3 cycles of a front-line taxane and platinum-containing regimen prior to entry on this study.
5. Patients must have a documented complete clinical response on front-line therapy.
6. Patients must be disease-free from prior malignancies for more than 5 years with the exception of curatively-treated basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix.
7. Life expectancy of > 6 months.
8. ECOG (Zubrod) performance status 0-2.
9. Age >18 years.
10. Patient has the following blood counts at Baseline:

    * ANC > 1.5 x 10-9 c/L;
    * platelets > 100 x 10-9 c/L;
    * Hgb > 9 g/dL.
11. Patient has the following blood chemistry levels at Baseline:

    * AST (SGOT), ALT (SGPT) < 1.5x upper limit of normal range (ULN);
    * total bilirubin NORMAL;
    * alkaline phosphatase < 2.5x ULN
    * creatinine < 1.5 mg/dL.
12. Patient or his/her legally authorized representative or guardian has been informed about the nature of the study, and has agreed to participate in the study, and signed the Informed Consent form prior to participation in any study-related activities.

Exclusion Criteria:

1. Patients who have received more than one prior chemotherapy regimen.
2. Evidence of active brain metastases, including leptomeningeal involvement. Prior evidence of brain metastasis permitted only if treated and stable off therapy for at least 1 month.
3. Patient has pre-existing peripheral neuropathy of grade >/= 2 (per National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events version 3.0 [CTCAE].
4. Patients receiving concurrent or intervening other chemotherapy, hormonal (for treatment of ovarian carcinoma), immunotherapy, or radiotherapy.
5. Patient has a clinically significant concurrent illness.
6. Patient is, in the Investigator's opinion, unlikely to be able to complete the study through the End of Study (EOS) visit.
7. Patient has a history of allergy or hypersensitivity to the study drug.
8. Patient has serious medical risk factors involving any of the major organ systems such that the investigator considers it unsafe for the patient to receive an experimental research drug.
9. Patient is enrolled in any other clinical protocol or investigational trial.
10. Patients of childbearing potential, not practicing adequate contraception.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2005-11; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Response Rate | 5 years

SECONDARY OUTCOMES:
Time to Response | 5 years
Duration of Response | 5 years
Overall Survival | 5 years
Progression Free Survival | 5 years
Safety | 5 years
Tolerability | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Benidict B Benigno, MD, Principal Investigator — Southeastern Gynecologic Oncology
Locations (1):
- Southeastern Gynecologic Oncology, Atlanta, Georgia, United States